CLINICAL TRIAL: NCT06424171
Title: Atrial Fibrillation and the Risk of Stroke in Veteran athLETES: a Pilot Cardiac and Cerebral Magnetic Resonance Imaging Study - AFLETES-MRI
Brief Title: AFLETES-MRI: A Cardiac and Cerebral Magnetic Resonance Imaging Study in Athletes With Atrial Fibrillation
Acronym: AFLETES-MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0917
Record Dates: First submitted 2024-02-26; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Athletes with atrial fibrillation without diagnosed stroke.
  Interventions: Diagnostic Test: Cardiac and brain magnetic resonance imaging.
- Athletes without atrial fibrillation.
  Interventions: Diagnostic Test: Cardiac and brain magnetic resonance imaging.
- Athletes with atrial fibrillation and a diagnosed stroke.
  Interventions: Diagnostic Test: Cardiac and brain magnetic resonance imaging.
- Healthy, non-athlete controls.
  Interventions: Diagnostic Test: Cardiac and brain magnetic resonance imaging.

INTERVENTIONS:
Diagnostic Test: Cardiac and brain magnetic resonance imaging. — Cardiac magnetic resonance imaging with analysis using 4D flow. Brain magnetic resonance imaging to detect strokes, including microvascular strokes.

SUMMARY:
Participation in exercise improves cardiovascular health. However, long-term endurance exercise may increase the risk of an irregular heart rhythm called atrial fibrillation (AF).

In AF, blood flow is altered, increasing the risk of clot formation in the heart which may enter the circulation and cause a stroke. The risk of stroke can be reduced with the use of blood thinning medication. Athletes with atrial fibrillation, due to their healthy lifestyle, are generally felt to be at low risk of stroke and many would not be offered blood thinning treatment using risk scores used in clinical practice.

In a recent survey of almost one thousand athletes, the investigators found that there was an increased risk of stroke in those with atrial fibrillation, even in those without other risk factors for stroke.

To further investigate these findings, this study will use MRI scanning to look at the hearts and brains of athletes aged between 40-64 years old. The researchers will assess athletes with and without atrial fibrillation, as well as some athletes with atrial fibrillation who have had a stroke previously.

The MRI scans will measure heart size and function as well as blood flow patterns in the heart. The study will determine whether athletes with atrial fibrillation have evidence of stroke on brain MRI and whether these are related to abnormal flow patterns. The results will help us decide whether a larger study should be performed.

ELIGIBILITY:
Inclusion Criteria:

* Male, atrial fibrillation.
* 40-64 years of age at the time of enrolment.
* Primarily (≥50% of competition) competes in an endurance type sport as defined by European Society of Cardiology 2020 guidelines.
* Competitive athlete*
* CHA2-DS2-VAsc =0/1 (excluding previous stroke).

  * Competitive athlete defined by having trained ≥10 years, 6 hours per week as a self-reported average and having participated in at least one competitive event at regional level or above.

Exclusion Criteria:

* History of pre-existing cardiovascular disease
* Previous myocardial infarction, peripheral arterial disease
* Left ventricular systolic dysfunction (EF <45%)
* Heart muscle disease
* Complex congenital heart disease.
* Moderate or severe valvular disease.
* Uncontrolled hypertension (180/100mmHg)
* Clotting or bleeding disorders, vasculitis
* Inherited cerebral disease
* Known to have an estimated glomerular filtration rate <30 ml/min/1.73m2.

Ages: 40 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: - Male, competitive, veteran athletes and age/sex matched controls will be included.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Stroke. | Baseline.
  The number of participants with ischaemic white matter lesions, micro-infarcts and old infarcts.

SECONDARY OUTCOMES:
Cardiac structure. | Baseline.
  Left ventricular volume (ml).
Late gadolinium enhancement (LGE). | Baseline.
  Presence of LGE. The number of participants with LGE will be compared between groups.
Left atrial flow-pathlines and streamlines. | Baseline.
  Direction of pathlines and streamlines. The number of areas of stasis will be calculated for each group.
Cardiac function. | Baseline.
  Ejection fraction of the left ventricular (%).
Left atrial stasis. | Baseline.
  Number of areas of stasis in each group in the left atrium.

CONTACTS AND LOCATIONS:
Overall Officials: Gerry P McCann, MD, MRCP(UK), MB,ChB, Study Chair — University of Leicester; Susil Pallikadavath, MRCP(UK), MBChB(hons), BSc, Principal Investigator — University of Leicester
Locations (1):
- Department of Cardiovascular Sciences, University of Leicester, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Background] Newman W, Parry-Williams G, Wiles J, Edwards J, Hulbert S, Kipourou K, Papadakis M, Sharma R, O'Driscoll J. Risk of atrial fibrillation in athletes: a systematic review and meta-analysis. Br J Sports Med. 2021 Nov;55(21):1233-1238. doi: 10.1136/bjsports-2021-103994. Epub 2021 Jul 12. PMID 34253538
- [Background] Pallikadavath S, Richards C, Bountziouka V, Sandilands AJ, Graham-Brown MPM, Robinson T, Singh A, McCann GP. The AFLETES Study: Atrial Fibrillation in Veteran Athletes and the Risk of Stroke. Clin J Sport Med. 2023 May 1;33(3):209-216. doi: 10.1097/JSM.0000000000001115. Epub 2023 Apr 6. PMID 37042823
- [Background] Dyverfeldt P, Bissell M, Barker AJ, Bolger AF, Carlhall CJ, Ebbers T, Francios CJ, Frydrychowicz A, Geiger J, Giese D, Hope MD, Kilner PJ, Kozerke S, Myerson S, Neubauer S, Wieben O, Markl M. 4D flow cardiovascular magnetic resonance consensus statement. J Cardiovasc Magn Reson. 2015 Aug 10;17(1):72. doi: 10.1186/s12968-015-0174-5. PMID 26257141
- [Background] Lippi G, Sanchis-Gomar F, Cervellin G. Global epidemiology of atrial fibrillation: An increasing epidemic and public health challenge. Int J Stroke. 2021 Feb;16(2):217-221. doi: 10.1177/1747493019897870. Epub 2020 Jan 19. PMID 31955707
- [Background] Xu Y, Zhao L, Zhang L, Han Y, Wang P, Yu S. Left Atrial Enlargement and the Risk of Stroke: A Meta-Analysis of Prospective Cohort Studies. Front Neurol. 2020 Feb 14;11:26. doi: 10.3389/fneur.2020.00026. eCollection 2020. PMID 32117002
- [Background] Androulakis E, Swoboda PP. The Role of Cardiovascular Magnetic Resonance in Sports Cardiology; Current Utility and Future Perspectives. Curr Treat Options Cardiovasc Med. 2018 Aug 31;20(10):86. doi: 10.1007/s11936-018-0679-y. PMID 30167977
- [Background] Graham-Brown MP, Gulsin GS, Parke K, Wormleighton J, Lai FY, Athithan L, Arnold JR, Burton JO, McCann GP, Singh AS. A comparison of the reproducibility of two cine-derived strain software programmes in disease states. Eur J Radiol. 2019 Apr;113:51-58. doi: 10.1016/j.ejrad.2019.01.026. Epub 2019 Jan 23. PMID 30927959
- [Background] D'Ascenzi F, Anselmi F, Focardi M, Mondillo S. Atrial Enlargement in the Athlete's Heart: Assessment of Atrial Function May Help Distinguish Adaptive from Pathologic Remodeling. J Am Soc Echocardiogr. 2018 Feb;31(2):148-157. doi: 10.1016/j.echo.2017.11.009. Epub 2017 Dec 13. PMID 29246514
- [Background] Androulakis E, Mouselimis D, Tsarouchas A, Antonopoulos A, Bakogiannis C, Papagkikas P, Vlachopoulos C. The Role of Cardiovascular Magnetic Resonance Imaging in the Assessment of Myocardial Fibrosis in Young and Veteran Athletes: Insights From a Meta-Analysis. Front Cardiovasc Med. 2021 Dec 21;8:784474. doi: 10.3389/fcvm.2021.784474. eCollection 2021. PMID 34993239
- [Background] Demirkiran A, van Ooij P, Westenberg JJM, Hofman MBM, van Assen HC, Schoonmade LJ, Asim U, Blanken CPS, Nederveen AJ, van Rossum AC, Gotte MJW. Clinical intra-cardiac 4D flow CMR: acquisition, analysis, and clinical applications. Eur Heart J Cardiovasc Imaging. 2022 Jan 24;23(2):154-165. doi: 10.1093/ehjci/jeab112. PMID 34143872
- [Background] Suwa K, Saitoh T, Takehara Y, Sano M, Nobuhara M, Saotome M, Urushida T, Katoh H, Satoh H, Sugiyama M, Wakayama T, Alley M, Sakahara H, Hayashi H. Characteristics of intra-left atrial flow dynamics and factors affecting formation of the vortex flow - analysis with phase-resolved 3-dimensional cine phase contrast magnetic resonance imaging. Circ J. 2015;79(1):144-52. doi: 10.1253/circj.CJ-14-0562. Epub 2014 Nov 13. PMID 25391258
- [Background] Fluckiger JU, Goldberger JJ, Lee DC, Ng J, Lee R, Goyal A, Markl M. Left atrial flow velocity distribution and flow coherence using four-dimensional FLOW MRI: a pilot study investigating the impact of age and Pre- and Postintervention atrial fibrillation on atrial hemodynamics. J Magn Reson Imaging. 2013 Sep;38(3):580-7. doi: 10.1002/jmri.23994. Epub 2013 Jan 4. PMID 23292793
- [Background] Lee DC, Markl M, Ng J, Carr M, Benefield B, Carr JC, Goldberger JJ. Three-dimensional left atrial blood flow characteristics in patients with atrial fibrillation assessed by 4D flow CMR. Eur Heart J Cardiovasc Imaging. 2016 Nov;17(11):1259-1268. doi: 10.1093/ehjci/jev304. Epub 2015 Nov 20. PMID 26590397
- [Background] Pelliccia A, Sharma S, Gati S, Back M, Borjesson M, Caselli S, Collet JP, Corrado D, Drezner JA, Halle M, Hansen D, Heidbuchel H, Myers J, Niebauer J, Papadakis M, Piepoli MF, Prescott E, Roos-Hesselink JW, Graham Stuart A, Taylor RS, Thompson PD, Tiberi M, Vanhees L, Wilhelm M; ESC Scientific Document Group. 2020 ESC Guidelines on sports cardiology and exercise in patients with cardiovascular disease. Eur Heart J. 2021 Jan 1;42(1):17-96. doi: 10.1093/eurheartj/ehaa605. No abstract available. PMID 32860412